CLINICAL TRIAL: NCT03188133
Title: Top Down Visual Information Processing in Schizophrenia Patients With Visual Hallucinations
Brief Title: Visual Information Processing in Schizophrenia Patients With Visual Hallucinations
Acronym: SHALL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ID-RCB/2017-A01058-45
Record Dates: First submitted 2017-06-09; First posted 2017-06-15 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Schizophrenia; Visual Hallucination; Auditory Hallucination; False Perception
Keywords: Schizophrenia; Visual Hallucination; False Perception; emotional priming
MeSH Terms: conditions — Schizophrenia; Hallucinations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VH (Experimental): schizophrenia patients with visual hallucinations
  Interventions: Other: behavioral task : emotional priming
- AH/NH (Active Comparator): schizophrenia patients with auditory hallucinations or no hallucinations
  Interventions: Other: behavioral task : emotional priming
- C (Active Comparator): healthy controls
  Interventions: Other: behavioral task : emotional priming

INTERVENTIONS:
Other: behavioral task : emotional priming — emotional priming task on ambiguous visual stimuli

SUMMARY:
Occurrence of visual hallucinations (VHs) in schizophrenia depend in part on disorders in the processing of late visual information (Top-Down). The broader question of how these top-down mechanisms (cognitive and / or emotional mechanisms) are involved in the occurrence of VHs remains to be specified and very few behavioral studies have so far been interested. The investigators propose to study the implication of Top-Down mechanisms in the visual hallucinatory manifestations, more specifically in the processing of ambiguous stimuli during an emotional priming task. Schizophrenia patients with VHs would have more false visual perceptions in the treatment of ambiguous stimuli than schizophrenia patients with auditory hallucinations or no hallucinations (AH/NH) and healthy controls.

DETAILED DESCRIPTION:
In schizophrenia patients with auditory hallucinations, top-down mechanism on perceptual processing could be illustrated by tasks of listening to white noise. These studies show that psychotic subjects detect more words and phrases when exposed to these stimuli. In schizophrenia patients with VHs, to our knowledge no study have explored the mechanism of false perception. Thus, we propose to experimentally manipulate the implication of Top-Down mechanisms on visual perception using an emotional priming task. This paradigm has already been used in this population to explain the mechanisms underlying productive symptoms. For example, in an emotional priming task authors have shown that a negative valence primer contributes to the implementation of an interpretive bias in a confidence judgment task.

The aim of the present study is to explore the implication of these Top-Down mechanisms in hallucinatory manifestations, more specifically on the treatment of ambiguous visual stimuli during an emotional priming task by manipulating the emotional valence of the primer. The goal is to determine how emotional environmental elements contribute to the formation of erroneous perceptions in patients with schizophrenia with VHs.

ELIGIBILITY:
All Groups:

* Age between 18 and 55 years
* Affiliation to or benefiting from a social security
* Visual acuity normal or corrected to normal
* Person who received and understood the complete information about the organization of the research and gave written and free informed consent before participating in the study

Group of patients with schizophrenia with visual hallucination (HV) with or without auditory hallucination (HA) (HV group):

* Schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders IV criteria
* Presence of a hallucinatory visual symptomatology (HV) in the history of the disease measured by the Psychosensory hallucination scale (PSAS).
* The presence of a hallucinatory symptomatology in auditory mode (HA) in addition to the HV is not a criterion of non-inclusion.

Group of patients with schizophrenia either with auditory hallucination (HA) but without visual hallucination (HV) or no hallucination, auditory or visual (NH) (HA / NH group)

* Schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders IV criteria
* Presence of a hallucinatory symptomatology in auditory mode (HA) in the history of the disease measured by the PSAS or absence of any hallucinatory manifestations in the history of the disease
* Absence of visual hallucinatory symptomatology (HV) in the history of the disease as measured by PSAS

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-10-17 (Estimated); Primary Completion 2018-05-01 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of false visual perception on the emotional priming task | through study completion an average of 6 months
  Number of false perception made by participants on an ambiguous visual stimulus i.e when a participant identifies incorrectly an ambiguous stimulus as a genuine percept (for example a participant sees a face in a noisy grey pattern)

SECONDARY OUTCOMES:
number of false visual perception on the emotional priming task depending of the emotional valence manipulated | through study completion an average of 6 months
  The investigators will investigate if the manipulated valence of the emotional priming task influences the number of false visual perceptions of ambiguous stimuli
Cognitive performances at the neuropsychological assessment | through study completion an average of 6 months
  Cognitive performances at the neuropsychological assessment conducted for both groups of schizophrenia patients. Neuropsychological assessment will provide performance scores on different cognitive functions : episodic memory (California Verbal Learning Test), visual memory (delayed match to sample task), working memory (forward and backward digit span, n-back task), sustained attention (test of attentional performance battery), divided attention (test of attentional performance battery), inhibition (test of attentional performance battery), processing speed (coding) and visual perception and processing (visual object space perception task).
Psychosensory hallucinations scale scores | through study completion an average of 6 months
  scores on the Psychosensory hallucinations scale conducted for both schizophrenia patients groups. This scale provides a complete evaluation of hallucinations in all modalities as well as the impact of these symptoms on daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent LAPREVOTE, Principal Investigator — Central hospital Nancy, Centre Psychothérapique de Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catalan A, Simons CJ, Bustamante S, Drukker M, Madrazo A, de Artaza MG, Gorostiza I, van Os J, Gonzalez-Torres MA. Novel evidence that attributing affectively salient signal to random noise is associated with psychosis. PLoS One. 2014 Jul 14;9(7):e102520. doi: 10.1371/journal.pone.0102520. eCollection 2014. PMID 25020079
- [Background] Hoffman RE, Woods SW, Hawkins KA, Pittman B, Tohen M, Preda A, Breier A, Glist J, Addington J, Perkins DO, McGlashan TH. Extracting spurious messages from noise and risk of schizophrenia-spectrum disorders in a prodromal population. Br J Psychiatry. 2007 Oct;191:355-6. doi: 10.1192/bjp.bp.106.031195. PMID 17906248
- [Background] Galdos M, Simons C, Fernandez-Rivas A, Wichers M, Peralta C, Lataster T, Amer G, Myin-Germeys I, Allardyce J, Gonzalez-Torres MA, van Os J. Affectively salient meaning in random noise: a task sensitive to psychosis liability. Schizophr Bull. 2011 Nov;37(6):1179-86. doi: 10.1093/schbul/sbq029. Epub 2010 Apr 1. PMID 20360211
- [Background] Hooker CI, Tully LM, Verosky SC, Fisher M, Holland C, Vinogradov S. Can I trust you? Negative affective priming influences social judgments in schizophrenia. J Abnorm Psychol. 2011 Feb;120(1):98-107. doi: 10.1037/a0020630. PMID 20919787